CLINICAL TRIAL: NCT03990896
Title: Evaluation of Talazoparib, a PARP Inhibitor, in Patients With Somatic BRCA Mutant Metastatic Breast Cancer: Genotyping Based Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Neelima Vidula, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-188
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Talazoparib (Experimental): -Talazoparib will be provided as capsules for oral administration daily
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — Talazoparib is a study drug that inhibits (stops) the normal activity of certain proteins called "poly (ADP-ribose) polymerases" also called "PARPs". PARPs are proteins (made from genes which are part of DNA) that are found in all normal and cancer cells that are involved in the repair of DNA. PARPs are needed to repair mistakes that can happen in DNA when cells divide. If the mistakes are not repaired, the defective cell will usually die and be replaced. Cells with mistakes in their DNA that do not die can become cancer cells.
  Other Names: Talzenna

SUMMARY:
This research is to evaluate the effectiveness of Talazoparib as a potential treatment for metastatic breast cancer with a BRCA 1 or BRCA 2 mutation.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved talazoparib for the participants' specific disease but it has been approved for metastatic breast cancer with a germline (inherited) BRCA mutation.

Talazoparib is a study drug that inhibits (stops) the normal activity of certain proteins called "poly (ADP-ribose) polymerases" also called "PARPs". PARPs are proteins (made from genes which are part of your DNA) that are found in all normal and cancer cells that are involved in the repair of DNA. PARPs are needed to repair mistakes that can happen in DNA when cells divide. If the mistakes are not repaired, the defective cell will usually die and be replaced. Cells with mistakes in their DNA that do not die can become cancer cells. Cancer cells may be killed by a study drug, like talazoparib, that stops the normal activity of PARPs. In clinical trials, the use of talazoparib and other PARP inhibitors have shown that these drugs can reduce tumor size and slow tumor growth in some cancer patients with BRCA1 or BRCA2 mutations.

In this research study, the investigators are examining how effective talazoparib is in patients with metastatic breast cancer with a BRCA mutation in their tumor.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer with deleterious somatic BRCA 1 or 2 mutations detectable by cell-free circulating tumor DNA, by CLIA certified clinical assay (including but not restricted to MGH-Snapshot cfDNA assay, Guardant360, Foundation One). The eligibility of a given assay and/or BRCA mutation could be discussed with the primary investigator (Dr. Vidula) and senior investigator (Dr. Bardia), who will provide the final discretion.
* Patients with germline BRCA 1 or 2 mutations will not be eligible.
* Patients with only a VUS (Variant of Unknown Significance), or non-functional BRCA mutation, without a deleterious somatic BRCA 1 or 2 mutation will not be eligible.
* The following disease subtypes are eligible:

  * Triple negative breast cancer (defined as ER < 1%, PR < 1%, HER2 negative, as per ASCO CAP guidelines), with disease progression on at least one prior chemotherapy regimen in the metastatic setting.
  * Hormone receptor positive, HER2 negative disease with disease progression on at least one prior endocrine therapy in the metastatic setting or be considered inappropriate for endocrine therapy
* Patients must have evaluable or measurable disease.
* Any number of prior lines of therapy are allowed
* Patients may have received prior platinum based chemotherapy (0-1 prior platinum based therapy). However, the patient must not have progressed while on platinum treatment (any setting), or within 6 months after end of treatment (neoadjuvant and/or adjuvant).
* At least two weeks from last systemic therapy for breast cancer, with recovery of all treatment related toxicity to grade 1 or less. Subjects with ≤ Grade 2 neuropathy are an exception to this criterion.
* At least two weeks from last radiation therapy, with recovery of all treatment related toxicity to grade 1 or less.

  -≥ 18 years of age on day of signing informed consent.
* ECOG performance status of ≤2.
* Adequate organ function as defined in Table 1 within 10 days prior to treatment initiation.
* Adequate Organ Function Laboratory Values
* SYSTEM LABORATORY VALUE
* Hematological

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
* Renal

  --Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X institutional upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Hepatic

  * Serum total bilirubin ≤ 1.5 X institutional ULN OR Direct bilirubin ≤ institutional ULN for subjects with total bilirubin levels > 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X institutional ULN OR ≤ 5 X institutional ULN for subjects with liver metastases
* Prior CNS disease is allowed if stable for at least one month since whole brain radiation therapy in patients who received whole brain radiation, or 2 weeks since stereotactic radiotherapy in patients who received stereotactic radiotherapy. Patients should not be requiring steroids. Patients whose CNS disease was surgically treated may be enrolled if stable for at least one month after surgery, and not requiring steroids.
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must use an acceptable form of birth control per treating physician discretion or be surgically sterile, or abstain from heterosexual activity for the course of the study through 7 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy. Additionally, male patients may not donate sperm during the duration of the study and through 7 months after the last dose of study therapy.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Treatment with an investigational agent within 4 weeks of the first dose of treatment.
* Patients must not have received prior treatment with a PARP inhibitor
* Patients must not have a germline BRCA 1 or 2 mutation
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion.

  --If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known, untreated central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 7 months after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or Hepatitis C.
* Patients should not be on strong P-glycoprotein inhibitors.
* Patients should not be on any other anti-cancer therapy (chemotherapy, hormone therapy, immunotherapy, or alternate investigational therapy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Median Progression Free Survival | From the start of treatment until death or disease progression, up to approximately 2 years
  Progression-Free Survival (PFS) is defined as the time from the first dose of study treatment to the date of disease progression as assessed by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) or death due to any cause, whichever occurs first. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).

SECONDARY OUTCOMES:
Objective Response Rate | From the start of treatment until treatment discontinuation, up to approximately 2 years
  The number of participants that achieve either a complete (CR) or partial response (PR) according to RECIST 1.1.
  * CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Number of Participants with Treatment-related Serious Adverse Events | From the start of treatment until treatment discontinuation, up to approximately 2 years
  Adverse events will be assessed using Common Terminology Criteria for Adverse Events (CTCAE 5). The number of participants with grade 3 or greater adverse events that were deemed to be possibly, probably, or definitely related to study treatment will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Neelima Vidula, MD, Principal Investigator — Massachusetts General Hospital
Locations (7):
- United States (7):
  - UCSF Medical Center-Mission Bay/Benioff Children's Hospital, San Francisco, California
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Weill Cornell Medicine, New York, New York
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation